CLINICAL TRIAL: NCT02772757
Title: Efficacy of a Coupler-Based Hearing-Aid Fitting Approach for Experienced Users
Brief Title: Coupler-Based Hearing-Aid Fitting Approach for Experienced Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1895-P
Record Dates: First submitted 2016-05-02; First posted 2016-05-13 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-02

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aids; outcome assessment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care group (Active Comparator): Standard of Care group will receive the standard, face-to-face hearing aid fitting and verification approach
  Interventions: Behavioral: standard hearing aid fitting
- Average RECD group (Experimental): This group will have their hearing aid fitting via the coupler using average RECD values during the fitting
  Interventions: Behavioral: coupler-based fitting
- Measured RECD group (Experimental): This group will have their hearing aid fitting via the coupler using measured RECD values during the fitting
  Interventions: Behavioral: coupler-based fitting

INTERVENTIONS:
Behavioral: standard hearing aid fitting — standard hearing aid, face-to-face fitting
  Arms: Standard of Care group
Behavioral: coupler-based fitting — coupler-based fitting using average RECDs
  Arms: Average RECD group
Behavioral: coupler-based fitting — coupler-based fitting using measured RECDs
  Arms: Measured RECD group

SUMMARY:
The overall aim of the study is to compare the verification accuracy and hearing-aid outcomes between the traditional, fitting approach where the patient is present during the visit and a coupler-based fitting approach where the patient is not present and mailed their hearing aids. If the coupler-based fitting protocol tested in this study as effective as the traditional fitting protocol, then patients receiving replacement hearing aids may circumvent a face-to-face visit.

DETAILED DESCRIPTION:
This study will incorporate a verification technique that simulates the patient's actual ear during probe microphone verification measurements, called real-ear to coupler difference (RECD). Because the patient's ear is not used during the RECD measurement, but rather simulated, the patient would not need to be present during the RECD verification. This RECD hearing aid verification can occur in the clinic after which the hearing aids will be mailed to the patient. This study will compare the fitting accuracy and outcomes between the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* no more than a moderate sensorineural hearing loss (defined as < 60 dB HL pure-tone average at 500, 1000, and 2000 Hz AU)
* experienced BTE hearing-aid users who are obtaining replacement VA-issued BTE hearing aids coupled to a custom earmold that is simply an upgrade in model with the same style earmold
* ability to read and write in English as determined by reading a few sentences from the consent document aloud so that self-report measures can be completed

Exclusion Criteria:

* outer or middle ear pathology as determined by otoscopy, immittance, and/or audiometric testing (e.g., conductive or mixed losses)
* lack of phone or non-use of the phone as the participants will be required to conduct a telephone interview after they obtain their replacement hearing aids
* unwilling or unable to be mailed hearing aids
* co-morbid condition that would preclude their participation as determined by a chart review

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherri L Smith, PhD, Principal Investigator — Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN
Locations (1):
- Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN, Mountain Home, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Click here for more information about this study: Efficacy of a Coupler-Based Hearing-Aid Fitting Approach for Experienced Users — http://www.avreap.research.va.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Experienced hearing-aid users were recruited from the Mountain Home VA Audiology Clinic in Mountain Home, TN
Pre-assignment Details: A total of 77 participants were consented. A total of 5 participants did not meet the inclusion criteria and thus were not randomized because they didn't qualify. A total of 72 participants were randomized.
Period: Overall Study
Arm/Group | Standard of Care Group | Average RECD Group | Measured RECD Group
Started | 22 | 24 | 26
Completed | 21 | 21 | 21
Not Completed | 1 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Physician Decision | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Group | Average RECD Group | Measured RECD Group | Total
Number analyzed (Participants) | 21 | 21 | 21 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.24 (6.13) | 71.24 (6.05) | 72.57 (4.97) | 72.02 (5.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 21 | 21 | 21 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 21 | 21 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 19 | 19 | 20 | 58
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 21 | 63

OUTCOME MEASURES:

1. Primary Outcome: in Situ Real-ear Aided Response (REAR)
Description: Deviation from prescriptive target (re: in situ REAR) from both ears of each participant for each group. This measure reflects the accuracy of the hearing aid fittings from 250 Hz through 3000 Hz (the average bandwidth of audibility).
Time Frame: at the visit where in-situ real ear measurements are made (immediate post-fitting)
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Standard of Care Group | Average RECD Group | Measured RECD Group
Number analyzed (Participants) | 21 | 21 | 21
dB | -.21 (0.80) | -1.86 (2.95) | 0.05 (2.36)

2. Secondary Outcome: Client-Oriented Scale of Improvement (COSI)
Description: The listener nominates up to five listening goals. After hearing-aid use, the listener assesses two outcomes for each goal. One outcome is the degree of change relative to the patient's unaided experience. Responses are recorded on a 5 unit categorical scale from 'worse' to 'much better'. The second outcome is the final satisfactory 'aided' ability for each goal as measured on a 5 unit categorical scale from hardy ever (10%) to almost always (95%). Higher scores reflect better outcomes for nominated goals. We calculated the percent of better and much better responses over the nominated goals and the average satisfactory aided ability over the nominated goals.
Time Frame: 1 month post-fitting
Population: One participant in the Average RECD group and one participant in the Measured RECD group declined to nominate listening goals and complete the measure. Two additional participants in the Measured RECD group did not wear the replacement hearing aids due to comfort and thus did not complete self-report measures related to the field trial.
Measure: Mean (Standard Deviation); unit: percentage of change or ability
Arm/Group | Standard of Care Group | Average RECD Group | Measured RECD Group
Number analyzed (Participants) | 21 | 20 | 18
percentage of change or ability
  degree of change | 87.3 (26.3) | 82.9 (30.2) | 71.8 (36.5)
  final ability | 78.2 (15.2) | 80.0 (20.8) | 67.8 (27.2)

3. Secondary Outcome: Device Oriented Subjective Outcome (DOSO) Scale
Description: The questionnaire is comprised of 28 items making up the following six subscales related to listening performance with hearing aids: (1) speech cues, (2) listening effort, (3) pleasantness, (4) quietness, (5) convenience, and (6) use. Responses from 'not at all' (1 point) to tremendously (7 points) are recorded for each item and are averaged across all items to obtain a total scale score. Higher scores reflect higher outcomes. The minimum and maximum total scores can range from 1-7 and for the three groups were: standard of care group (3.8-6.8), Average RECD group (3.3-6.7), and measured RCD group (3.8-6.5).
Time Frame: 1 month post-fitting
Population: Two participants in the Measured RECD group did not wear the replacement hearing aids due to comfort and thus did not complete self-report measures related to the field trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care Group | Average RECD Group | Measured RECD Group
Number analyzed (Participants) | 21 | 21 | 19
units on a scale | 5.7 (0.8) | 5.9 (0.8) | 5.5 (0.7)

4. Secondary Outcome: Satisfaction With Amplification in Daily Life (SADL)
Description: The SADL questionnaire has 15 items that examine self-reported hearing-aid satisfaction. The following four subscales are included: (1) positive effect, (2) negative features, (3) personal image, and (4) service and cost. Item 14 is omitted in populations who do not pay for hearing aids. Responses are on a 1 to 7 scale with higher numbers reflecting higher outcomes. The item responses are averaged to determine the total satisfaction score that can range from 1-7. The minimum and maximum total scores for the three groups were: standard of care group (5.1-7.0); average RECD group (4.2-6.9), and measured RECD group (4.9-7.0).
Time Frame: 1 month post-fitting
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard of Care Group: This group received the standard of care fitting with in site real ear verification
Arm/Group | Standard of Care Group | Average RECD Group | Measured RECD Group
Number analyzed (Participants) | 21 | 21 | 19
units on a scale | 6.2 (0.6) | 6.0 (0.6) | 6.0 (0.5)

ADVERSE EVENTS:
Time Frame: 1 year and 3 months
Description: Our definition of adverse events is the same as clinical trials.gov.
Arm/Group | Standard of Care Group | Average RECD Group | Measured RECD Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
Pilot study limited to one style of hearing aids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT02772757/Prot_SAP_000.pdf